CLINICAL TRIAL: NCT00263523
Title: PET Imaging of Brain 5-HT1A Receptors Using [11C](-)-RWAY
Brief Title: PET Imaging of Brain 5-HT(1A) Receptors Using [(11)C](-)-RWAY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060042; 06-M-0042
Record Dates: First submitted 2005-12-08; First posted 2005-12-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-15

CONDITIONS: Healthy Volunteers
Keywords: Serotonin; Positron Emission Tomograhy; Brain; Neurochemistry; Neurotransmitter; Healthy Volunteer; HV
MeSH Terms: interventions — 2, 3, 4, 5, 6, 7-hexahydro-1(4-(1(4-(2-methoxyphenyl)-piperazinyl))-2-phenylbutyry)-1H-azepine

INTERVENTIONS:
Drug: [11C] (-)-RWAY

SUMMARY:
This study will use positron emission tomography (PET) and magnetic resonance imaging (MRI) to measure a serotonin receptor subtype in the brain called 5-HT(1A). This receptor is a target for drug therapy to treat anxiety and depression. The study will see if a newly developed radioligand (radioactive substance used in PET scanning to study the receptor systems of the brain) called [(11)C](-)-RWAY is more effective than other radioligands currently used in brain receptor research.

Healthy subjects 18-40 years of age may be eligible for this study. Candidates are screened with a physical examination, electrocardiogram, and blood and urine tests.

Participants undergo PET and MRI scanning as follows:

PET scan

PET uses small amounts of a radioactive chemical called a tracer (in this case, [(11)C](-)-RWAY) that "labels" active areas of the brain. For the procedure, the subject lies on the scanner bed. A special mask is fitted to the subject's head and attached to the bed to help keep the head still during the scan so the images will be clear. A brief scan is done just before the tracer is injected to provide measures of the brain that will help in the precise calculation of information from subsequent scans. Then, the tracer is injected through a catheter (plastic tube) placed in the arm and pictures are taken for about 2 hours, while the subject lies still on the scanner bed. Subjects return to the clinic for blood and urine tests 24 hours after the scan.

MRI

The MRI scan is done within 1 year of the PET scan. MRI uses a magnetic field and radio waves to produce images of body tissues and organs-in this case, the brain. The subject lies on a table that is moved into the scanner (a tube-like device), wearing earplugs to muffle the noise of the machine during the scanning process. The space in the scanner is confining and may cause some people to be somewhat anxious. An intercom system allows the subject to speak with the staff member performing the study at all times during the procedure, and the procedure can be stopped at any time.

DETAILED DESCRIPTION:
The 5-hydroxytryptamine (serotonin, 5-HT) 5-HT(1A) receptors subtype is a target for drug therapy in the treatment of anxiety and depression. Radioligands currently in use with PET for studying human brain 5-HT(1A) receptors in clinical research or drug development are based on WAY-100635. Though variously effective, they each suffer from one or more drawbacks with respect to measuring relative regional receptor densities. These drawbacks include: rapid metabolism and very low non-specific binding for [carbonyl-(11)C]WAY-100635; defluoridation for [18F]trans-FCWAY. Therefore, we have recently developed [(11)C](-)-RWAY as an alternative radioligand for brain 5 HT(1A) receptors. Even though similar to WAY-100635, [(11)C](-)-RWAY has a reversed amide linkage. Reversal of the direction of the amide bond may confer resistance to amide hydrolysis and make acceptable easy labeling at its O-methoxy group. In the present protocol, we plan to perform a kinetic brain imaging study in healthy human subjects to measure 5 HT(1A) receptors in brain regions with [(11)C](-)-RWAY.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must be healthy and aged 18-65 years.

EXCLUSION CRITERIA:

Current psychiatric illness, substance abuse or severe systemic disease based on history and physical exam.

Any existing physical exam and ECG within one year will be reviewed and if none already exists in the chart, these will be obtained and reviewed.

Laboratory tests with clinically significant abnormalities.

Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual limits.

Pregnancy and breast feeding.

Claustrophobia.

Presence of ferromagnetic metal in the body or heart pacemaker.

Positive HIV test.

A history of brain disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-12-05; Study Completion 2007-08-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Burger C, Buck A. Requirements and implementation of a flexible kinetic modeling tool. J Nucl Med. 1997 Nov;38(11):1818-23. PMID 9374364